CLINICAL TRIAL: NCT06508554
Title: The Door to the Womb at Birth: Haptonomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Burcu KUCUKKAYA, Assist. Prof, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2023-SBB-0594
Record Dates: First submitted 2024-07-13; First posted 2024-07-18 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Birth Outcome, Adverse; Self Efficacy; Memory Impairment; Pregnancy Related
Keywords: Haptonomy; Birth Expectation
MeSH Terms: conditions — Pregnancy Complications; Memory Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No action will be taken. Surveys and scales will be applied.
- Haptonomy (Experimental): 1. A face-to-face sitting position will be taken for the application.
  2. Throughout the research, the study will be accompanied by the music desired by each pregnant woman. The same music chosen by the woman or couple will be used throughout the work.
  3. The application will be done with the pregnant woman's eyes closed.
  4. The application will start with breathing exercises and the body will be relaxed with the help of abdominal and chest breathing (hara breathing).
  5. With the energy work, we will move on to the stage of harmonizing the intuitive and heart energy fields. The researcher and the pregnant woman will place their left hands on each other's hearts. The aim is to feel the energy flowing from each other, to feel the heart, to open the third eye and to prepare the hands. This study aims to increase the pregnant woman's confidence in her own emotions and body by getting to know her emotions and body.
  Interventions: Other: Haptonomy

INTERVENTIONS:
Other: Haptonomy — 5. With the energy work, we will move on to the stage of harmonizing the intuitive and heart energy fields. It will be ensured that the mother's communication with her baby has a spiritual dimension as well as a physical one. 6. Then the stage of touching and communicating with the baby will begin. The hands of the researcher and the pregnant woman will be placed on the pregnant woman's uterus. Then, the pregnant woman will be the first to call her baby. This call to the baby will be repeated 2-3 times. 7. The pregnant woman and her uterus will be touched and exercises will be performed to adapt to the fetus. The aim is to increase the emotional awareness of the pregnant woman and to enable her to play intrauterine games with her baby (such as calling the baby, shaking her belly, moving the baby to the touched area with the mother's voice). Haptonomy will be completed with a deep relaxation exercise that will support the heart-uterus connection accompanied by breathing exercises.
  Arms: Haptonomy

SUMMARY:
Purpose: This study aimed to examine the effect of haptonomy application on the expectant mother's birth expectations, experiences, birth self-efficacy, birth memory and reminder during labor.

Materials and Methods: The prospective, double-blind, randomized controlled study is conducted between 10.10.2023-10.08.2024, with n=80 (40=control, 40=intervention) women volunteering to participate in the study randomly in two groups: intervention and control. In the study, the Personal Data Collection Form prepared by reviewing the literature, Wijma Birth Expectation/Experience Scale (W-DEQ) A and B version, Labor Self-Efficacy Scale (DEÖÖ) and Birth Memory and Recall Scale (DHÖ) were used.

ELIGIBILITY:
Inclusion Criteria:

* Married and pregnant women,
* ≥ 18 years old,
* Able to read, write and understand Turkish,
* Living in the city center where the study is conducted,
* Does not have any physical or psychological health problems for herself or her baby,
* Having a spontaneous pregnancy at 28.< gestational weeks,
* Those who have not received haptonomy application before,
* Pregnant women who agreed to participate in the study were included.

Exclusion Criteria:

* Those with psychological and chronic health problems,
* Pregnant women who did not agree to participate in the study were not included.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-02-25 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Wijma Birth Expectation/Experience Scale (W-DEQ) A and B version | change before the application of the patent and after the 32nd, 34th, 36th, 38th weeks of pregnancy and the 1st day and 1st month postpartum.
  This scale was adapted from Wijma et al. Developed by. The purpose of the scale is to evaluate women's fear of birth during their own birth experiences in the postpartum period. Turkish validity and reliability study was conducted by Uçar and Beji. The scale consists of 33 items. Each item is a 6-point Likert type with scores ranging from 1 to 6, with 1 being "completely" and 6 being "not at all". While the minimum score on the scale is 33, the maximum score is 198. High scores indicate that women have a high fear of childbirth. Negatively loaded questions in the scale (2, 3, 6, 7, 8, 11, 12,15, 19, 20, 24, 25, 27, 31) are calculated by reversing them in the opposite direction to ensure consistency in measurement.
Self-Efficacy Scale in Labor | change before the application of the patent and after the 32nd, 34th, 36th, 38th weeks of pregnancy and the 1st day and 1st month postpartum.
  Self-Efficacy Scale in Labor - Short Version' was developed by Ip et al. to measure self-efficacy levels in labor. The Turkish validity and reliability study of the scale was conducted by Ersoy (2011). The scale consists of two sub-dimensions: outcome expectation and competence expectation, and there are 16 questions in each sub-dimension. The lowest score to be obtained from the sub-dimensions of the scale is 16 and the highest score is 160. A high score from each subscale indicates that pregnant women have high expectations of adequacy and outcome regarding labor. Responses on a Likert-type scale are scored from 1 to 10.
Birth Memory and Recall Scale | change before the application of the patent and after the 32nd, 34th, 36th, 38th weeks of pregnancy and the 1st day and 1st month postpartum.
  This scale developed by Foley et al. in 2014, was adapted into Turkish by Topkara and Çağan in 2021. The scale is a 7-point Likert type. The scale, which consists of a total of 21 items, has six sub-dimensions. Its sub-dimensions are "Emotional Memory", "Ambivalent Emotional Memory", "Centeredness of Memory", "Coherence and Reliving", "Sensory Memory" and "Involuntary Remembering". The highest score that can be obtained from the scale is 147 and the lowest score is 6. High scores from the "Emotional Memory" sub-dimension indicate that the mother's negative emotions about the birth experience are more intense, high scores from the "Ambivalent Emotional Memory" sub-dimension indicate that the mother has more ambivalent emotions, and high scores from the "Centeredness of Memory" sub-dimension indicate that the mother has more ambivalent emotions.

CONTACTS AND LOCATIONS:
Locations (1):
- Bartın University, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided